CLINICAL TRIAL: NCT06124703
Title: Comparing Two Dosing Regimens of the Efficacy of Short-term Oral Prednisone Therapy on Acute Subjective Tinnitus
Brief Title: Different Dosing Regimens of STOP-AST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: different STOP-AST regimens
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss; Tinnitus; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss; Tinnitus; Hearing Loss, Sensorineural | interventions — Prednisone; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose-tapering regimen (Active Comparator): The dose selection of oral prednisone is the maximum daily dose for 4 days, followed by a taper every 2 days
  Interventions: Drug: Prednisone tablet; Drug: Ginkgo Biloba Extract
- no taper regimen (Experimental): The dose selection of oral prednisone is the maximum daily dose, applied for 5 consecutive days
  Interventions: Drug: Prednisone tablet; Drug: Ginkgo Biloba Extract

INTERVENTIONS:
Drug: Prednisone tablet — Prednisone acetate tablet (5 mg prednisone acetate per tablet) was provided
  Other Names: Prednisone
Drug: Ginkgo Biloba Extract — Ginkgo biloba extract (EGb) is a compound drug derived from Ginkgo biloba trees native to China.
  Other Names: EGb

SUMMARY:
The goal of this clinical trial is to learn about the different dose regimens of the efficacy of oral steroids in the acute tinnitus population. Participants will receive different appropriate dosages of prednisone tablets and oral Ginkgo Biloba tablets.

DETAILED DESCRIPTION:
The purpose of this clinical study was to investigate the efficacy and to compare two different oral doses of short-term systemic steroid therapy for acute tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old;
2. primary complaint of subjective tinnitus ≤ 1 months of duration;
3. a decline in auditory function by audiological assessments on the day of the test, of which the outcome must either satisfy one of the following conditions:

   1. a reduced distortion product otoacoustic emissions (DPOAE) amplitude in individuals with normal Pure tone audiometry (PTA) results;
   2. more than a PTA threshold > 20 dB with frequencies between 125 and 8000 Hz, but not exhibited idiopathic sudden sensorineural hearing loss;
4. a state of good general condition;
5. with good adherence to participation and signed informed consent.

Exclusion Criteria:

1. active middle ear pathology;
2. patients who had received treatment for their current condition prior to the study;
3. both the PTA and DPOAE with normal outcomes;
4. hearing implants;
5. history of known corticosteroids contraindications (including osteoporosis, peptic ulcers, poorly controlled hypertension, diabetes, chronic liver or renal insufficiency, tumorous condition, alcohol abuse, pregnant patients, and women on estrogen-containing oral contraceptive steroids).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
tinnitus handicap inventory (THI) | one week from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus
tinnitus handicap inventory (THI) | two weeks from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus
tinnitus handicap inventory (THI) | one month from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus

SECONDARY OUTCOMES:
visual analog scale (VAS) | one week from baseline
  mark the severity of tinnitus on a horizontal scale from 0 to 10. The higher the score, the more severe the symptoms.
visual analog scale (VAS) | two weeks from baseline
  mark the severity of tinnitus on a horizontal scale from 0 to 10. The higher the score, the more severe the symptoms.
visual analog scale (VAS) | one month from baseline
  mark the severity of tinnitus on a horizontal scale from 0 to 10. The higher the score, the more severe the symptoms.
the Athens Insomnia Scale-8 (AIS-8) | one week from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
the Athens Insomnia Scale-8 (AIS-8) | two weeks from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
the Athens Insomnia Scale-8 (AIS-8) | one month from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).

CONTACTS AND LOCATIONS:
Overall Officials: Shan Sun, Principal Investigator — Eye and ENT Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No